CLINICAL TRIAL: NCT05877222
Title: A Single-center, Open-label, Randomized, Crossover Phase 1 Trial to Investigate Bioequivalence Between 5 × 10 mg Tablets and 2 × 25 mg Tablets of Daridorexant in Healthy Male and Female Japanese Participants
Brief Title: A Phase 1 Trial to Investigate the Biological Equivalence of 5 × 10 mg Tablets and 2 × 25 mg Tablets of Daridorexant in Healthy Male and Female Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ID-078-127
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (5 × 10 mg daridorexant) (Experimental): Participants will receive a single oral dose of 5 × 10 mg daridorexant.
  Interventions: Drug: Daridorexant 10 mg
- Treatment B (5 × 25 mg daridorexant) (Experimental): Participants will receive a single oral dose of 2 × 25 mg daridorexant.
  Interventions: Drug: Daridorexant 25 mg

INTERVENTIONS:
Drug: Daridorexant 10 mg — Daridorexant will be available as film-coated tablets for oral administration formulated at strengths of 10 mg.
  Arms: Treatment A (5 × 10 mg daridorexant)
Drug: Daridorexant 25 mg — Daridorexant will be available as film-coated tablets for oral administration formulated at strengths of 25 mg.
  Arms: Treatment B (5 × 25 mg daridorexant)

SUMMARY:
A Phase 1 trial to investigate bioequivalence between 5 × 10 mg tablets and 2 × 25 mg tablets of daridorexant in healthy male and female Japanese participants

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any trial-mandated procedure.
* Healthy male and female participants aged between 18 and 65 years (inclusive) at Screening.
* Body mass index of 18.5 to 29.9 kg/m2 (inclusive) at Screening.
* Participant must be of native Japanese descent (all parents/grandparents of Japanese descent).
* Participant must not have been away from Japan for more than 10 years (at Screening visit).
* Participant's lifestyle should not have changed significantly since relocation from Japan.

Exclusion Criteria:

* Known hypersensitivity to daridorexant, or any of its excipients.
* History of narcolepsy or cataplexy.
* Clinically relevant findings on the physical examination at Screening.
* Clinically relevant findings on 12-lead ECG, recorded after 5 min in a supine position at Screening.
* Clinically relevant findings in clinical laboratory tests (hematology and clinical chemistry) at Screening.
* Clinically relevant findings in systolic blood pressure, diastolic blood pressure, and pulse rate, measured on either arm, after 5 min in the supine position at Screening.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed if performed > 12 weeks prior to administration of first study treatment, cholecystectomy not allowed).
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood samples for PK analysis will be taken at several timepoints from treatment administration on Day 1 to Day 3 of Study periods 1 and 2 (Total duration: up to 4 days)
AUC0-t | Blood samples for PK analysis will be taken at several timepoints from treatment administration on Day 1 to Day 3 of Study periods 1 and 2 (Total duration: up to 4 days)

OTHER OUTCOMES:
Tmax | Blood samples for PK analysis will be taken at several timepoints from treatment administration on Day 1 to Day 3 of Study periods 1 and 2 (Total duration: up to 4 days)
AUC0-inf | Blood samples for PK analysis will be taken at several timepoints from treatment administration on Day 1 to Day 3 of Study periods 1 and 2 (Total duration: up to 4 days)
λz | Blood samples for PK analysis will be taken at several timepoints from treatment administration on Day 1 to Day 3 of Study periods 1 and 2 (Total duration: up to 4 days)
T1/2 | Blood samples for PK analysis will be taken at several timepoints from treatment administration on Day 1 to Day 3 of Study periods 1 and 2 (Total duration: up to 4 days)
Treatment-emergent AEs | From study treatment administration up to End-of-Treatment (EOT) (Total duration: up to 46 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Study Director, Study Director — Idosia Pharmaceuticals Ltd
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No